CLINICAL TRIAL: NCT03199079
Title: Cervix Monitor for Risk Assessment of Spontaneous Preterm Delivery
Brief Title: Cervix Monitor for Elasticity and Length Measurements
Status: Completed | Type: Observational
Sponsor: Advanced Tactile Imaging, Inc. (Industry)
Collaborators: Princeton Urogynecology (Other); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: CM01A/B
Record Dates: First submitted 2017-05-22; First posted 2017-06-26 (Actual); Results first posted 2020-04-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2020-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Group 1: Non-pregnant women: Non-pregnant women with normal pelvic floor
  Interventions: Other: Measurement
- Group 2: Pregnant women: Pregnant women; 22-29 weeks of pregnancy
  Interventions: Other: Measurement

INTERVENTIONS:
Other: Measurement — Measurement of cervix elasticity and length measurements is not an intervention

SUMMARY:
Preterm birth is a leading global cause of neonatal mortality despite of numerous advances and intensive research in perinatal medicine. Almost one million children die each year due to complications of preterm birth and in almost all countries with reliable data, preterm birth rates are increasing. Of the 14 million survivors per year, many face a lifetime of disability, including learning disabilities, visual and hearing impairments. Spontaneous preterm delivery (SPTD) is often multi factorial event, precocious cervical softening, shortening and dilatation are a common denominator. The majority of preterm births happen spontaneously, though some are due to early induction of labor or cesarean birth, typically due to medical maternal of neonatal conditions.

DETAILED DESCRIPTION:
The uterine cervix has to provide structural integrity and mechanical resistance to ensure normal development of the fetus as the uterus expands to accommodate the fetus growth. Preterm delivery is closely related to a premature cervical ripening. The scientific bases for the proposed project is the elasticity modulus of a cervix is a more sensitive parameter characterizing the stage of cervical ripening. The main component of the cervix tissue is a collagen. Cervical ripening is the result of realignment of collagen, degradation of collagen cross-linking due to proteolytic enzymes. These processes affect the elasticity modulus of the cervical tissue. Therefore, assessment of cervix by a device measuring cervical elasticity and cervical length appears to be and adequate approach for identifying pregnant women at high risk of spontaneous preterm delivery. The primary cervical elasticity assessment currently used in clinical practice is relying on the evaluation of the cervix as "hard, medium or soft". In the scope of this project the investigators propose to develop and clinically validate a new and cost-effective device, Cervix Monitor for detecting cervix conditions leading to SPTD and its risk assessment. The CM will be based on measuring of the applied pressure to the cervix by a tactile sensor array and ultrasound measurement of cervix length .

ELIGIBILITY:
Inclusion Criteria:

1. Adult women age 21-44 years
2. Non-pregnant women, or
3. Pregnant women

Exclusion Criteria:

1. Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder
2. Ongoing or prior radiation therapy for abdominal or pelvic cancer
3. Recent (less than four months) pelvic surgery
4. Surgically absent uterus, rectum or bladder
5. Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician
6. Severe abdominal or pelvic adhesions preventing access to pertinent anatomy
7. Known or suspected bleeding disorder
8. HIV or hepatitis B positive serology
9. Warty lesions on the vulva
10. Extensive varicose veins on the vulva
11. Active skin infection or ulceration within the vagina/vulva (Herpes infection)
12. Presence of a vaginal septum
13. Severe hemorrhoids

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult women
Study Population: Conditions precluding patients from participation are listed in the study exclusion criteria below. In addition, cognitively impaired patients will not be asked to participate. No patients will be excluded on the basis of race.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, PhD, Principal Investigator — Advanced Tactile Imaging, Inc.
Locations (2):
- United States (2):
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Princeton Urogynecology, Princeton, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Egorov V, Rosen T, van Raalte H, Kurtenoks V. Cervical Characterization with Tactile-Ultrasound Probe. Open J Obstet Gynecol. 2020 Jan;10(1):85-99. doi: 10.4236/ojog.2020.101008. Epub 2020 Jan 8. PMID 32133244

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-pregnant Women: Adult women age 21-44 years; 10 non-pregnant women
- Pregnant Women: Adult woman age 21-44 years; 22-29 weeks of pregnancy; 10 women
Period: Overall Study
Arm/Group | Non-pregnant Women | Pregnant Women
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Non-pregnant Women: Non-pregnant women with normal pelvic floor
  Cervix Monitor: Cervix elasticity and length measurements by Cervix Monitor
- Group 2: Pregnant Women: Pregnant women; 22-29 weeks of pregnancy
  Cervix Monitor: Cervix elasticity and length measurements by Cervix Monitor
- Total: Total of all reporting groups
Arm/Group | Group 1: Non-pregnant Women | Group 2: Pregnant Women | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (7.1) | 32.4 (5.6) | 34.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cervix Elasticity
Description: Young's modulus of the cervix at 4 locations. Units of measurement is kPa.
Time Frame: During examination procedure
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Non-pregnant Women | Pregnant Women
Number analyzed (Participants) | 10 | 10
kPa | 54 (17) | 19.7 (15.4)

2. Secondary Outcome: Cervix Length
Description: Cervix length in mm
Time Frame: During examination procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Non-pregnant Women | Pregnant Women
Number analyzed (Participants) | 10 | 10
mm | 42 (13) | 30.7 (6.6)

ADVERSE EVENTS:
Time Frame: Nine (9) months
Description: Cervix monitor device is a low risk device. All-Cause Mortality was not monitored/assessed.
Arm/Group | Non-pregnant Women | Pregnant Women
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03199079/Prot_SAP_000.pdf